CLINICAL TRIAL: NCT06357754
Title: Protocol for Transgene Assay Service
Brief Title: Transgene Assay Testing Service of Tumor Samples From Patients Who Received a Bristol-Myers Squibb Manufactured Gene Modified Cell Therapy and Have a Qualifying Second Primary Malignancy
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA082-085
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukaemia; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Multiple Myeloma | interventions — idecabtagene vicleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Acceptable sample types for transgene testing include:
  * Formalin fixed paraffin embedded (FFPE) tumor sample (twenty 4-5 μm freshly cut sections)
  * Bone marrow aspirate (up to 6mL. minimum of 4mL)
  * FFPE bone marrow biopsy (twenty 4-5 μm freshly cut sections)
  * Peripheral blood (6ml)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated with idecabtagene vicleucel
  Interventions: Biological: Idecabtagene vicleucel
- Participants treated with lisocabtagene maraleucel
  Interventions: Biological: Lisocabtagene maraleucel

INTERVENTIONS:
Biological: Idecabtagene vicleucel — As per product label
  Groups: Participants treated with idecabtagene vicleucel
Biological: Lisocabtagene maraleucel — As per product label
  Groups: Participants treated with lisocabtagene maraleucel

SUMMARY:
The purpose of this transgene assay testing service is to evaluate tumor samples for transgene levels in patients who received a commercially available Bristol-Myers Squibb manufactured gene modified cellular therapy and have reported a qualifying second malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has received a commercially available Bristol-Myers Squibb (BMS) manufactured Gene Modified Cell Therapy (GMCT) and has been diagnosed with a qualifying second primary malignancy or a second primary malignancy which BMS has qualified for testing.
* Participant has received a commercially available BMS manufactured GMCT in a clinical trial or other investigational setting (including non-conforming product) for which there is no testing protocol in place for that trial or investigational setting and has been diagnosed with a qualifying second primary malignancy or a second primary malignancy which BMS has qualified for testing.

Exclusion Criteria:

* Participant is actively participating in a clinical trial where information and sample collection is being conducted under that clinical trial.
* Participant has not received a BMS manufactured GMCT or has not been diagnosed with a qualifying second primary malignancy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants who receive a Bristol-Myers Squibb (BMS) manufactured Gene Modified Cell Therapy (GMCT) that have been diagnosed with a qualifying secondary malignancy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2038-10-06 (Estimated); Study Completion 2038-10-06 (Estimated)

PRIMARY OUTCOMES:
Participant in situ hybridization (ISH) or droplet-based digital Polymerase chain reaction (ddPCR) transgene testing results | Baseline
Participant insertion site analysis (ISA) testing results | Baseline
  For participants with positive in situ hybridization (ISH) transgene or droplet-based digital polymerase chain reaction (ddPCR) transgene

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (4):
  - Local Institution - 0016, Portland, Oregon
  - Ut Southwestern, Dallas, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Local Institution - 0004, Madison, Wisconsin
- Universitaetsklinikum Essen (AoR), Essen, Germany
- Japan (2):
  - Toyokawa City Hospital, Toyokawa, Aichi-ken
  - Local Institution - 0003, Kumamoto, Kumamoto
- Kantonsspital Aarau, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts